CLINICAL TRIAL: NCT02113267
Title: Treatment of Eosinophilic Esophagitis With Mometason Furoat Aerosol: a Randomised, Placebo-controled Phase II Study for Evaluation of Treatment Effect on Group Level Including Symtom Questionnaires
Brief Title: Mometasone-furoate for Treatment of Eosinophilic Esophagitis - a Randomized Placebo Controlled Study.
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Combination slow recruitment, short shelf life for placebo and insufficient funding for further drug production (probably anyway sufficient number included).
Sponsor: Mogens Bove (Other Government)
Collaborators: Vastra Gotaland Region (Other Government)
Responsible Party: Sponsor-Investigator, Mogens Bove, Associate Professor, Vastra Gotaland Region
Organization: Vastra Gotaland Region (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VGFOUREG-226361; 2012-005842-39 (EudraCT Number)
Record Dates: First submitted 2014-04-10; First posted 2014-04-14 (Estimated); Last update posted 2018-10-17 (Actual); Status verified 2018-10

CONDITIONS: Eosinophilic Esophagitis
Keywords: esophagitis; eosinophils; allergy; inflammation; corticosteroids
MeSH Terms: conditions — Eosinophilic Esophagitis; Esophagitis; Hypersensitivity; Inflammation | interventions — Mometasone Furoate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Mometasone furoat (Experimental): Mometasone furoate monohydrate. 4 spray doses à 50 micrograms by mouth to be swallowed 4 times daily after meals (9) with no eating or drinking allowed 30 minutes after intake. Duration of treatment is 8 weeks.
  Interventions: Drug: Mometasone furoate
- Placebo spray (Placebo Comparator): Placebo. 4 spray doses à 50 micrograms by mouth to be swallowed 4 times daily after meals (9) with no eating or drinking allowed 30 minutes after intake. Duration of treatment is 8 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Mometasone furoate — 4 spray doses à 50 micrograms by mouth to be swallowed 4 times daily after meals with no eating or drinking allowed 30 minutes after intake. Duration of treatment is 8 weeks.
  Other Names: Nasonex
  Arms: Mometasone furoat
Drug: Placebo — 4 spray doses à 50 micrograms by mouth to be swallowed 4 times daily after meals (9) with no eating or drinking allowed 30 minutes after intake. Duration of treatment is 8 weeks.
  Other Names: Nasonex comparator spray (APL)
  Arms: Placebo spray

SUMMARY:
Background:

Eosinophilic esophagitis ( EoE ) is a disease entity which has been properly recognized only within the past two decades.(1) A prevalence of nearly 1% means that almost 20,000 people in the Region of Western Sweden may be affected.(2 ) The main symptom is swallowing difficulty and food may be stuck, which typically require acute hospital care with operational action under general anesthesia.( 3,4 ) The standard treatment today is local treatment with steroids by mouth several times a day for a few weeks.( 5 ) In adults and large teenagers, there is only one randomized study which has shown that budesonide has a significant effect exaggerating that of placebo. However, the main end-point in this study was the degree of tissue inflammation.(6) In a separate study using validated questionnaires , we have shown that patients with EoE have distinct organ-specific symptoms and a lowered quality of life . These symptoms nearly disappeared, after treatment with mometasone furoate. However, as that study was not randomized or placebo controlled no causal conclusions could be drawn regarding the treatment effect, but the method of validated questionnaires proved sensitive to changes in symptomatology.(7) Purpose The primary purpose of this study is to evaluate the effect of local steroid treatment with mometasone furoate on swallowing problems in patients with EoE . Secondarily, to evaluate the effect on patient quality of life and the presence of side effects.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years
* Newly diagnosed cases with diagnostic criteria for EoE (ie at least 15 eosinophils per high power field (Magnification 10 times 40 = x400) in any field of view in any esophageal biopsy and concurrent symptoms of esophageal dysfunction mainly dysphagia.
* Women of childbearing age may participate provided that the pregnancy is not planned , and that contraceptive use during therapy. The investigator will arrange a free pregnancy test must be performed within 1 week before treatment and be negative.
* Participation requires oral and written informed and signed consent form (see patient information and consent forms).

Exclusion Criteria:

* Local infection of the pharynx or esophagus , such as fungal, bacterial or viral infection
* Active or latent tuberculosis in respiratory tract
* Recent history of major trauma or major surgery
* Recent significant infection or other physical stress
* Signs or suspicion of dehydration
* History of injury, illness or surgery in the adrenals or pituitary
* Pharynx or esophagussurgery or other trauma in the esophagus (incl. foreign body with a sharp object ) where healing has not taken place. (in case of doubt to be assessed by esophago - gastroscopy.
* Planned elective surgery during treatment
* Pregnancy, ongoing or planned
* Women of childbearing potential not using preventives during the study period
* Glaucoma
* Hypersensitivity to any component in the treatments
* Systemic or local steroid treatment last 4 months
* Contraindication to steroid therapy ( immune deficiency or suppression , stomach ulcers, diabetes)
* Medications that affect oesophageal motility (cisapride, erythromycin ) during the treatment period .
* PPIs during or up to 2 weeks before the treatment period
* Other cause of dysphagia (cancer, connective tissue disease , neurological disease )
* Volunteer who can not consent to the study or complete a questionnaire

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2014-04 (Actual); Primary Completion 2018-09 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
Watson Dysphagia Scale Score (WDS) | Two months
  Difference in WDS score during treatment in active as compared to placebo group.

SECONDARY OUTCOMES:
The EORTC QLQ-OES18 dysphagia scale, the eating scale and choking item | Two months
  Difference in score in active- as compared to placebo- group

OTHER OUTCOMES:
"global health and social functioning dimensions" of SF-36 | Two months
  Difference in global health during treatment in active- as compared to placebo group.

CONTACTS AND LOCATIONS:
Overall Officials: Mogens Bove, MD,PhD, Principal Investigator — Dept of ENT, Head&Neck Surgery, NÄL Hospital, Trollhättan, Sweden
Locations (1):
- ENT dept, NÄL Hospital, Trollhättan, Sweden

REFERENCES:
- [Background] Bergquist H, Bove M. Eosinophilic esophagitis in adults: An ear, nose, and throat perspective. Laryngoscope. 2009 Aug;119(8):1467-71. doi: 10.1002/lary.20255. PMID 19504557
- [Background] Ronkainen J, Talley NJ, Aro P, Storskrubb T, Johansson SE, Lind T, Bolling-Sternevald E, Vieth M, Stolte M, Walker MM, Agreus L. Prevalence of oesophageal eosinophils and eosinophilic oesophagitis in adults: the population-based Kalixanda study. Gut. 2007 May;56(5):615-20. doi: 10.1136/gut.2006.107714. Epub 2006 Nov 29. PMID 17135307
- [Background] Larsson H, Bergquist H, Bove M. The incidence of esophageal bolus impaction: is there a seasonal variation? Otolaryngol Head Neck Surg. 2011 Feb;144(2):186-90. doi: 10.1177/0194599810392655. PMID 21493413
- [Background] Kerlin P, Jones D, Remedios M, Campbell C. Prevalence of eosinophilic esophagitis in adults with food bolus obstruction of the esophagus. J Clin Gastroenterol. 2007 Apr;41(4):356-61. doi: 10.1097/01.mcg.0000225590.08825.77. PMID 17413601
- [Background] Liacouras CA, Furuta GT, Hirano I, Atkins D, Attwood SE, Bonis PA, Burks AW, Chehade M, Collins MH, Dellon ES, Dohil R, Falk GW, Gonsalves N, Gupta SK, Katzka DA, Lucendo AJ, Markowitz JE, Noel RJ, Odze RD, Putnam PE, Richter JE, Romero Y, Ruchelli E, Sampson HA, Schoepfer A, Shaheen NJ, Sicherer SH, Spechler S, Spergel JM, Straumann A, Wershil BK, Rothenberg ME, Aceves SS. Eosinophilic esophagitis: updated consensus recommendations for children and adults. J Allergy Clin Immunol. 2011 Jul;128(1):3-20.e6; quiz 21-2. doi: 10.1016/j.jaci.2011.02.040. Epub 2011 Apr 7. PMID 21477849
- [Background] Straumann A, Conus S, Degen L, Felder S, Kummer M, Engel H, Bussmann C, Beglinger C, Schoepfer A, Simon HU. Budesonide is effective in adolescent and adult patients with active eosinophilic esophagitis. Gastroenterology. 2010 Nov;139(5):1526-37, 1537.e1. doi: 10.1053/j.gastro.2010.07.048. Epub 2010 Aug 1. PMID 20682320
- [Background] Bergquist H, Larsson H, Johansson L, Bove M. Dysphagia and quality of life may improve with mometasone treatment in patients with eosinophilic esophagitis: a pilot study. Otolaryngol Head Neck Surg. 2011 Oct;145(4):551-6. doi: 10.1177/0194599811409857. Epub 2011 May 18. PMID 21593463
- [Derived] Tytor J, Larsson H, Bove M, Johansson L, Bergquist H. Topically applied mometasone furoate improves dysphagia in adult eosinophilic esophagitis - results from a double-blind, randomized, placebo-controlled trial. Scand J Gastroenterol. 2021 Jun;56(6):629-634. doi: 10.1080/00365521.2021.1906314. Epub 2021 Apr 8. PMID 33831327